CLINICAL TRIAL: NCT06167460
Title: Analysis of Circulating Tumor DNA Dynamics to Predict and Monitor Response to Tyrosine Kinase Inhibitors in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Analysis of Circulating Tumor DNA Dynamics to Predict and Monitor Response to TKI in Patients With Advanced NSCLC.
Status: Recruiting | Type: Observational
Sponsor: Gene Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: GS_ZTKL
Record Dates: First submitted 2023-11-21; First posted 2023-12-12 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Non Small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IIIC Non-Small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer; Tyrosine Kinase Inhibitors
Keywords: Liquid Biopsy; Circulating Tumour DNA; Vietnam
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The 1st blood sample is collected from eligible participants of non-small cell lung cancer, stage IIIB-IV, before TKI and chemotherapy.
  The 2nd -8th blood sample are collected from the participants every 3 months during TKI treatment, 6-8 sections of formalin-fixed paraffin-embedded (FFPE) tumor samples before TKI and chemotherapy are also collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an observational study, aiming to investigate whether the ctDNA dynamics analyzed by the K-TrackTM assay could predict early response to Tyrosine kinase inhibitors (TKIs) in patients with advanced non-small cell lung cancer (NSCLC).

1. Determine relationship between ctDNA dynamics and clinical response to TKI,

   * No response/progressive disease = ctDNA levels increase from baseline
   * Partial response/stable disease = ctDNA levels decrease from baseline
   * Complete response = ctDNA clearance.
2. Compare and combine ctDNA dynamics and RECIST1.1 to predict clinical response.
3. Determine relationship between ctDNA dynamics and progression free survival, overall survival.

DETAILED DESCRIPTION:
This study is recruiting female and male patients, aged 18 and older:

* Who are diagnosed with advanced non-small cell lung cancer and indicated for TKI (first or second line). TKI combined with chemotherapy is allowed,
* Who have not started TKI / chemotherapy before enrollment,
* Who have no medical or psychiatric conditions or occupational responsibilities that may preclude compliance with the protocol,
* FFPE/FNA sample is available,
* Compliant with treatment protocol,
* Patients consented to participate in the study. As part of the protocol, demographic data, medical and family history, and any relevant prior concomitant medication data will be recorded during follow-up visits. All patients are to be followed for 2 years from enrollment, with CT scan imaging measured every clinical visit for 24 months.

Sample collection:

* 10 mL of peripheral blood (in Streck tubes) is collected for ctDNA analysis at 8 time points: pre-treatment (<10 days before TKI), during TKI every 3 months until 21 months.
* 6-8 sections of formalin-fixed paraffin-embedded (FFPE) tumor samples before TKI/chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients are diagnosed with advanced non-small cell lung cancer and indicated for TKI (first or second line). TKI combined with chemotherapy is allowed.
* FFPE/FNA sample is available.
* Compliant with treatment protocol.
* Patients consented to participate in the study.

Exclusion Criteria:

* Patients already started TKI before enrollment.
* Patients already started chemotherapy before enrollment.
* Medical or psychiatric conditions or occupational responsibilities that may preclude compliance with the protocol.
* Patients did not agree to participate in the studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study population will include female and male, aged 18 and older, who are diagnosed with stage IIIB-IV Non-small cell lung cancer and indicated for TKI or TKI combined with chemotherapy. Eligible participants will meet all of the inclusion and exclusion criteria to be recruited into this study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Relationship between ctDNA dynamics and clinical response to TKI | 24 months following up.
  * No response/progressive disease = ctDNA levels increase from baseline
  * Partial response/stable disease = ctDNA levels decrease from baseline
  * Complete response = ctDNA clearance.
To compare and combine ctDNA dynamics and RECIST1.1 to predict clinical response. | 24 months following up.
  * Correlation between ctDNA dynamics and clinical response
  * Correlation between RECIST1.1 and clinical response
  * Combination of ctDNA dynamics and RECIST v1.1 in the prognosis of clinical response.
To investigate the relationship between ctDNA dynamics and progression free survival, overall survival. | 24 months following up.
  * Correlation between ctDNA dynamics and PFS
  * Correlation between ctDNA dynamics and OS.

CONTACTS AND LOCATIONS:
Overall Officials: Sinh D Nguyen, PhD, Principal Investigator — MGI
Locations (1):
- Medical Genetics Institute, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data of this this study may be requested for publication by the journals, sharing anonymized data with suitable study will be decided by the sponsor, PIs and the authority agency where the data was collected. No identifiable information will be shared with any other person/organization than authority in the study.
Supporting Information: Study Protocol, ICF
Time Frame: December 2025.
Access Criteria: GS_ZTKL for non-small cell lung cancer.

REFERENCES:
- [Background] Yang J, Gong Y, Lam VK, Shi Y, Guan Y, Zhang Y, Ji L, Chen Y, Zhao Y, Qian F, Chen J, Li P, Zhang F, Wang J, Zhang X, Yang L, Kopetz S, Futreal PA, Zhang J, Yi X, Xia X, Yu P. Deep sequencing of circulating tumor DNA detects molecular residual disease and predicts recurrence in gastric cancer. Cell Death Dis. 2020 May 11;11(5):346. doi: 10.1038/s41419-020-2531-z. PMID 32393783
- [Background] Reinert T, Henriksen TV, Christensen E, Sharma S, Salari R, Sethi H, Knudsen M, Nordentoft I, Wu HT, Tin AS, Heilskov Rasmussen M, Vang S, Shchegrova S, Frydendahl Boll Johansen A, Srinivasan R, Assaf Z, Balcioglu M, Olson A, Dashner S, Hafez D, Navarro S, Goel S, Rabinowitz M, Billings P, Sigurjonsson S, Dyrskjot L, Swenerton R, Aleshin A, Laurberg S, Husted Madsen A, Kannerup AS, Stribolt K, Palmelund Krag S, Iversen LH, Gotschalck Sunesen K, Lin CJ, Zimmermann BG, Lindbjerg Andersen C. Analysis of Plasma Cell-Free DNA by Ultradeep Sequencing in Patients With Stages I to III Colorectal Cancer. JAMA Oncol. 2019 Aug 1;5(8):1124-1131. doi: 10.1001/jamaoncol.2019.0528. PMID 31070691
- [Background] Magbanua MJM, Swigart LB, Wu HT, Hirst GL, Yau C, Wolf DM, Tin A, Salari R, Shchegrova S, Pawar H, Delson AL, DeMichele A, Liu MC, Chien AJ, Tripathy D, Asare S, Lin CJ, Billings P, Aleshin A, Sethi H, Louie M, Zimmermann B, Esserman LJ, van 't Veer LJ. Circulating tumor DNA in neoadjuvant-treated breast cancer reflects response and survival. Ann Oncol. 2021 Feb;32(2):229-239. doi: 10.1016/j.annonc.2020.11.007. Epub 2020 Nov 21. PMID 33232761
- [Background] Christensen E, Birkenkamp-Demtroder K, Sethi H, Shchegrova S, Salari R, Nordentoft I, Wu HT, Knudsen M, Lamy P, Lindskrog SV, Taber A, Balcioglu M, Vang S, Assaf Z, Sharma S, Tin AS, Srinivasan R, Hafez D, Reinert T, Navarro S, Olson A, Ram R, Dashner S, Rabinowitz M, Billings P, Sigurjonsson S, Andersen CL, Swenerton R, Aleshin A, Zimmermann B, Agerbaek M, Lin CJ, Jensen JB, Dyrskjot L. Early Detection of Metastatic Relapse and Monitoring of Therapeutic Efficacy by Ultra-Deep Sequencing of Plasma Cell-Free DNA in Patients With Urothelial Bladder Carcinoma. J Clin Oncol. 2019 Jun 20;37(18):1547-1557. doi: 10.1200/JCO.18.02052. Epub 2019 May 6. PMID 31059311
- [Background] Coombes RC, Page K, Salari R, Hastings RK, Armstrong A, Ahmed S, Ali S, Cleator S, Kenny L, Stebbing J, Rutherford M, Sethi H, Boydell A, Swenerton R, Fernandez-Garcia D, Gleason KLT, Goddard K, Guttery DS, Assaf ZJ, Wu HT, Natarajan P, Moore DA, Primrose L, Dashner S, Tin AS, Balcioglu M, Srinivasan R, Shchegrova SV, Olson A, Hafez D, Billings P, Aleshin A, Rehman F, Toghill BJ, Hills A, Louie MC, Lin CJ, Zimmermann BG, Shaw JA. Personalized Detection of Circulating Tumor DNA Antedates Breast Cancer Metastatic Recurrence. Clin Cancer Res. 2019 Jul 15;25(14):4255-4263. doi: 10.1158/1078-0432.CCR-18-3663. Epub 2019 Apr 16. PMID 30992300
- [Background] Labgaa I, Villacorta-Martin C, D'Avola D, Craig AJ, von Felden J, Martins-Filho SN, Sia D, Stueck A, Ward SC, Fiel MI, Mahajan M, Tabrizian P, Thung SN, Ang C, Friedman SL, Llovet JM, Schwartz M, Villanueva A. A pilot study of ultra-deep targeted sequencing of plasma DNA identifies driver mutations in hepatocellular carcinoma. Oncogene. 2018 Jul;37(27):3740-3752. doi: 10.1038/s41388-018-0206-3. Epub 2018 Apr 9. PMID 29628508
- [Background] Nguyen HT, Nguyen TV, Nguyen Hoang VA, Tran DH, Le Trinh NA, Le MT, Nguyen Tran TA, Pham TH, Dinh TC, Nguyen TS, Nguyen The KC, Mai H, Chu MT, Pham DH, Nguyen XC, Ngo Ha TM, Nguyen DS, Nguyen DQ, Lu YT, Do Thi TT, Truong DK, Nguyen QT, Nguyen HN, Giang H, Tu LN. Tumor genomic profiling and personalized tracking of circulating tumor DNA in Vietnamese colorectal cancer patients. Front Oncol. 2022 Dec 12;12:1069296. doi: 10.3389/fonc.2022.1069296. eCollection 2022. PMID 36578946
- [Background] Nguyen Hoang VA, Nguyen ST, Nguyen TV, Pham TH, Doan PL, Nguyen Thi NT, Nguyen ML, Dinh TC, Pham DH, Nguyen NM, Nguyen DS, Nguyen DQ, Lu YT, Do TTT, Truong DK, Phan MD, Nguyen HN, Giang H, Tu LN. Genetic landscape and personalized tracking of tumor mutations in Vietnamese women with breast cancer. Mol Oncol. 2023 Apr;17(4):598-610. doi: 10.1002/1878-0261.13356. Epub 2023 Jan 15. PMID 36495126
- [Background] Wei YF, Huang WT, Liu TC, Shieh JM, Chian CF, Wu MF, Chang CC, Lin CH, Ko JC, Lin CM, Hsia TC. Factors associated with improvement in symptoms and quality of life for first-line EGFR-tyrosine kinase inhibitor treatment in patients with EGFR-mutated non-small-cell lung cancer - A multicenter prospective SMILE study. J Cancer. 2019 Jul 10;10(17):4151-4158. doi: 10.7150/jca.30507. eCollection 2019. PMID 31417660
- [Background] Michelotti A, de Scordilli M, Bertoli E, De Carlo E, Del Conte A, Bearz A. NSCLC as the Paradigm of Precision Medicine at Its Finest: The Rise of New Druggable Molecular Targets for Advanced Disease. Int J Mol Sci. 2022 Jun 17;23(12):6748. doi: 10.3390/ijms23126748. PMID 35743191
- [Background] Horn L, Whisenant JG, Wakelee H, Reckamp KL, Qiao H, Leal TA, Du L, Hernandez J, Huang V, Blumenschein GR, Waqar SN, Patel SP, Nieva J, Oxnard GR, Sanborn RE, Shaffer T, Garg K, Holzhausen A, Harrow K, Liang C, Lim LP, Li M, Lovly CM. Monitoring Therapeutic Response and Resistance: Analysis of Circulating Tumor DNA in Patients With ALK+ Lung Cancer. J Thorac Oncol. 2019 Nov;14(11):1901-1911. doi: 10.1016/j.jtho.2019.08.003. Epub 2019 Aug 22. PMID 31446141
- [Background] Tran HT, Lam VK, Elamin YY, Hong L, Colen R, Elshafeey NA, Hassan ISA, Altan M, Blumenschein GR, Rinsurongkawong W, Rivera MJ, Vasquez ME, Carter BW, Byers LE, Tsao AS, Gibbons DL, Fossella F, Glisson BS, Zhang J, Heymach JV. Clinical Outcomes in Non-Small-Cell Lung Cancer Patients Treated With EGFR-Tyrosine Kinase Inhibitors and Other Targeted Therapies Based on Tumor Versus Plasma Genomic Profiling. JCO Precis Oncol. 2021 Aug 5;5:PO.20.00532. doi: 10.1200/PO.20.00532. eCollection 2021 Aug. PMID 34377884
- [Background] Mack PC, Miao J, Redman MW, Moon J, Goldberg SB, Herbst RS, Melnick MA, Walther Z, Hirsch FR, Politi K, Kelly K, Gandara DR. Circulating Tumor DNA Kinetics Predict Progression-Free and Overall Survival in EGFR TKI-Treated Patients with EGFR-Mutant NSCLC (SWOG S1403). Clin Cancer Res. 2022 Sep 1;28(17):3752-3760. doi: 10.1158/1078-0432.CCR-22-0741. PMID 35713632
- [Background] Soo RA, Martini JF, van der Wekken AJ, Teraoka S, Ferrara R, Shaw AT, Shepard D, Calella AM, Polli A, Toffalorio F, Tomasini P, Chiu CH, Kowalski DM, Kim HR, Solomon BJ. Early Circulating Tumor DNA Dynamics and Efficacy of Lorlatinib in Patients With Treatment-Naive, Advanced, ALK-Positive NSCLC. J Thorac Oncol. 2023 Nov;18(11):1568-1580. doi: 10.1016/j.jtho.2023.05.021. Epub 2023 Jun 7. PMID 37295609
- [Background] Gray JE, Ahn MJ, Oxnard GR, Shepherd FA, Imamura F, Cheng Y, Okamoto I, Cho BC, Lin MC, Wu YL, Majem M, Gautschi O, Boyer M, Bulusu KC, Markovets A, Barrett JC, Hodge R, McKeown A, Hartmaier RJ, Chmielecki J, Papadimitrakopoulou VA, Ramalingam SS. Early Clearance of Plasma Epidermal Growth Factor Receptor Mutations as a Predictor of Outcome on Osimertinib in Advanced Non-Small Cell Lung Cancer; Exploratory Analysis from AURA3 and FLAURA. Clin Cancer Res. 2023 Sep 1;29(17):3340-3351. doi: 10.1158/1078-0432.CCR-22-3146. PMID 37379430